CLINICAL TRIAL: NCT04368299
Title: Use of Telemedicine for Follow-up of Systemic Lupus Erythematosus ("TeleSLE") in the COVID-19 Outbreak: a Pragmatic Randomised Controlled Trial
Brief Title: Telemedicine for Follow-up of Systemic Lupus Erythematosus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ho SO, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TeleSLE
Record Dates: First submitted 2020-04-25; First posted 2020-04-29 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: SLE
MeSH Terms: interventions — Telemedicine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine (Experimental): Telemedicine group will receive scheduled follow-ups via videoconferencing.
  Interventions: Other: Telemedicine
- Standard care (Active Comparator): Standard care group patients will continue conventional standard in-person outpatient care.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Telemedicine — Videoconferencing for follow-up
  Arms: Telemedicine
Other: Standard care — Standard in-person outpatient follow-up
  Arms: Standard care

SUMMARY:
Background Patients with systemic lupus erythematosus (SLE) might be more susceptible to Covid-19 due to the underlying disease, co-morbidities and the use of immunosuppressive drugs. The investigators hypothesize that telemedicine (TM) can be an effective mode of health-care delivery minimizing the risk of SARS-CoV-2 exposure, while maintaining disease control in these patients.

Objectives The primary aim of this study is to evaluate the effectiveness to achieve remission or lupus low disease activity state (LLDAS) using TM delivered care compared to conventional in-person outpatient follow-up in SLE. The secondary objectives are to compare the patient reported outcomes and cost between the two modes of health care delivery.

Study design This is a 12-months single centered pragmatic randomized controlled study. A total of 150 enrolled patients with SLE being followed at the Prince of Wales Hospital rheumatology clinics will be randomized to either TM (TM group) or standard care (SC group) in a 1:1 ratio. Patients in the TM group will receive scheduled follow-ups via videoconferencing using a custom-made mobile app. SC group patients will continue conventional standard in-person outpatient care. The disease and patient reported outcomes as well as the health care related costs will be compared.

Expected outcomes Data from this study will support the notion that TM based care is as effective as conventional in-person care in achieving disease remission or LLDAS, as well as addressing psychosocial implications to ensure the best possible care for our patients in a cost-effective manner during this pandemic.

DETAILED DESCRIPTION:
There is a single-center pragmatic randomized controlled trial over a 12-month period. The study will be performed at the Rheumatology clinics at the Prince of Wales Hospital, which is a regional hospital in Hong Kong.

From May to October 2020, all consecutive patients with a diagnosis of SLE according to the 2019 European League Against Rheumatism/American College of Rheumatology classification criteria will be invited to participate in the study if they are aged >18 years, able to speak or understand Chinese and are willing to come back for routine blood and urine tests [18]. Patients (or carers) need to possess the technology needed to conduct a TM visit - a smartphone, tablet, or computer. Patients will be excluded if they are pregnant or incapable of answering a questionnaire. Patients will be randomization to either TM (TM group) or standard follow-ups (SF group 1). Patients who refused to be randomized will be offered standard in-person outpatient follow-up (SF group 2). All patients who fulfill the inclusion criteria and have given written informed consent will be asked to complete the Systemic Lupus Activity Questionnaire (SLAQ), LupusPRO, Health Assessment Questionnaire Disability Index (HAQ-DI), Medical Outcomes Survey Short Form (SF-36), Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale (version 4) and Hospital Anxiety and Depression Scale (HADS). They will also be asked to rate the confidence to the mode of care on a 10-point Likert scale (0 = not at all confident to 10 = very much confident). Their demographic, socio-economic and clinical data will be collected. Patient will be randomized in a ratio of 1:1 to either TM group or SF group 1 using a computer-generated random number sequence.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfilling the 2019 European League Against Rheumatism/American College of Rheumatology classification criteria
2. Over 18 years of age
3. able to speak or understand Chinese
4. willing to come back for routine blood and urine tests
5. possess the technology needed to conduct a TM visit

Exclusion Criteria:

1. pregnant
2. incapable of answering a questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
The percentage of patients in remission or LLDAS at one year. | 1 year

SECONDARY OUTCOMES:
Direct and indirect costs after one year. | 1 year
The change of Lupus Quality of Life (LupusQoL) at one year. | 1 year
  LupusQoL evaluates 8 domains including physical health, pain, planning, intimate relationships, burden to others, emotional health, body image, and fatigue. Questionnaire has a 5-point Likert response format (0=all the time, 1=most of the time, 2=a good bit of the time, 3=occasionally, and 4=never). Higher score means better quality of life.
Patient confidence and satisfaction score at one year. | 1 year
  They are in a 5-point Likert response format (0=strongly disagree, 1=disagree, 2=neutral, 3=agree, and 4=strongly agree). Higher score means more confident and satisfied.
Rates of adverse reaction and severe adverse reaction, including contracting COVID-19 infection, after one year. | 1 year
Numbers of clinic visits, hospitalization, overall in-person hospital visits in one year. | 1 year
The change of (Health Assessment Questionnaire Disability Index HAQ-DI) at one year. | 1 year
  HAQ-DI covers various common daily activities to assess disability.It consists of 8 questions. Each question asks on a scale ranging from 0 to 3 if the categories can be performed without any difficulty (scale 0) up to cannot be done at all (scale 3). Higher score means higher disability.
The change of (Hospital Anxiety and Depression Scale) HADS at one year. | 1 year
  HADS was developed to assess anxiety and depression in medical patients. Each domain has 7 items. Each item are answered by the patient on a four point (0-3) response category so the possible scores ranged from 0 to 21 for anxiety and 0 to 21 for depression. Higher score means more likely the patient has anxiety or depression.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided